CLINICAL TRIAL: NCT05765656
Title: Evaluation of the Effectiveness of a Joint General Practitioner-Pharmacist Intervention on the Implementation of Benzodiazepine Deprescribing in the Elderly (BESTOPH-MG Trial): Protocol for a Cluster-randomized Controlled Trial
Brief Title: Effectiveness of a Joint General Practitioner-Pharmacist Intervention on Benzodiazepine Deprescribing in the Elderly
Acronym: BESTOPH-MG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nantes University Hospital (Other)
Collaborators: Université de Nantes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: RC21_0357
Record Dates: First submitted 2023-02-10; First posted 2023-03-13 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-02

CONDITIONS: Primary Care; Health Plan Implementation; Benzodiazepine Dependence; Elderly; Anxiety; Deprescribing
Keywords: Primary care; collaborative practice; health plan implementation; deprescribing; benzodiazepine; elderly
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Pragmatic cluster-randomized controlled trial
Masking Description: Non applicable
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GP - pharmacist collaboration and pharmacist motivational interviewing (Experimental): Once randomized, the patient will have three motivational interviews with their pharmacist. Each time, a report will be sent to the GP.
  Interventions: Behavioral: GP - pharmacist collaboration and pharmacist motivational interviewing
- Usual Care (No Intervention): The patient is handled by his GP and the pharmacist as usual (medical encounter plus medication dispensation)

INTERVENTIONS:
Behavioral: GP - pharmacist collaboration and pharmacist motivational interviewing — 1. Patients in the GP-CP clusters randomized to the intervention arm will be offered a joint GP-CP deprescribing intervention by their GP.
  2. After the encounter, the patients will go to the pharmacy to get their medication dispensed. They will be given education materials. The pharmacist will plan with the patients 3 Motivational Interviews which will address the risks of using BZDR, and the benefits and modalities of stopping them. The pharmacists will receive a 2-day training course in MI. They will be given guidelines on BZDR deprescribing. If required, the pharmacists will be supported in their first MI.
  3. Following each interview, the pharmacist will inform the GP by means of a formalized report of the points discussed. The pharmacist will inform the GP of the patient's choice or not to get involved in a deprescribing process and of the protocol followed. The objective of this exchange is to formalize the joint GP-CP intervention and to secure the deprescribing of BZDR.
  Arms: GP - pharmacist collaboration and pharmacist motivational interviewing

SUMMARY:
Benzodiazepines or related drug (BZDR) are consumed for hypnotic or anxiolytic purposes in most cases. The consequences of BZDR are multiple with an increased risk of daytime sedation, balance disorders leading to falls and fractures, cognitive disorders, road accidents and dementia. Given their comorbidities, physiological changes, and multiple medications, the elderly are more at risk of suffering from BZDR adverse events.

Interprofessional collaboration has shown efficacy in improving prescribing appropriateness and may affect patients outcomes positively. Morever, motivational interviews (MI) may reduce the extent of substance abuse compared to no intervention.

DETAILED DESCRIPTION:
According to a 2017 report from the French National Agency for the Safety of Medicines and Health Products (ANSM), 13.4% of the French population used a benzodiazepine or related drug (BZDR) at least once in 2015. These drugs are consumed for hypnotic or anxiolytic purposes in most cases. As per the recommendations, BZDR should not be prescribed for more than 28 days when for hypnotic use and for 8 to 12 weeks, including withdrawal, when for anxiolytic purpose. Indeed, these drugs have shown a real, but mediocre, short-term efficacy on anxiety and sleep disorders. Moreover, their long-term effectiveness is almost nil. However, the literature shows that nearly one patient out of six taking a BZDR is a long-term user and that the proportion of patients for whom the indication is questionable can reach 2/3. The consequences of BZDR are multiple with an increased risk of daytime sedation, balance disorders leading to falls and fractures, cognitive disorders, road accidents and dementia. Also, given their comorbidities, physiological changes, and multiple medications, the elderly are more at risk of suffering from BZDR adverse events, like falls, driving accidents, dementia or even death. The majority of patients are unaware of these potential risks and continue to use these medications over the long term. They overestimate the benefits of BZDR and underestimate their harmful effects. The consequences are substantial, both from a health and financial perspective.

At the national level, numerous actions have been taken by the health authorities to reduce the use of BZDR: information for health professionals, pictograms on drug boxes, recommendations by health authorities, incentive measures by the Health Insurance services, or else health surveillance and regulatory measures to control prescribing. However, despite these numerous initiatives, the consumption of BZDR remains too high, even emphasized by the pandemic, and their deprescribing is struggling to be implemented in real life. Literature showed that many levers can facilitate the implementation of actions for the proper use of drugs. Interprofessional collaboration has shown efficacy in improving prescribing appropriateness and may affect patients outcomes positively, as shown by many recent systematic reviews and meta-analysis. General practitioners (GPs) who do not feel fully capable of implementing actions to deprescribe BZDR if they have to rely solely on guidelines, and because of the lack of time to re-evaluate these treatments. Yet, current international deprescribing studies remain based on actions only directed at the prescriber. Collaboration between two primary care professionals therefore appears to be a solution for implementing a medical decision to stop treatment. In addition, GPs are faced with a population which is very often reluctant to stop for fear of a return of anxiety or insomnia. In this context, another lever usable to achieve the implementation of deprescribing is the use of techniques that allow the patient to accept the physician's intervention. As such, motivational interviews (MI) may reduce the extent of substance abuse compared to no intervention. Developing and promoting training for healthcare professionals in MI may be a simple and pragmatic implementation strategy to reduce BZDR use.

ELIGIBILITY:
Inclusion Criteria:

* outpatients aged 65 and over
* followed by the general practitioner and the pharmacist of the GP-PO pair
* having a prescription for an anxiolytic or hypnotic BZDR prescribed at least 4 times in the past year
* the last prescription being less than 3 months old
* having been dispensed monthly during the last 3 months
* affiliated to a social security scheme
* and having given consent to participate in the research.

Exclusion Criteria:

* patients living in an institution
* participating in a clinical trial
* with epilepsy
* active depression
* uncontrolled mental disorders
* unable to participate in an interview or answer a questionnaire (demented, non-French speaking, illiterate, deaf, ...)
* under guardianship
* with a dystonic syndrome
* and patients who are not sufficiently autonomous to carry out the steps inherent in the study

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-03-15 (Estimated); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
Appropriateness measured by sociological interviews of patients, general practicioners and pharmacists and pharmacists observations | 3 to 6 months after the beginning of the enrollment period and 12 months after the end of the enrollment period
  Four days of observations will be conducted with pharmacists who have just been trained in MI to study, in action, how they conduct their first interviews with the elderly. These same pharmacists will be observed a second time at the end of the study, to see how their approach to MI has evolved. A first wave of ten semi-structured interviews will be conducted with elderly patients who have already been seen by their pharmacist, to see what effects the pharmacist has had on their representations of BZDR and on their consumption. Finally, three focus groups will be carried out, one with CPs, one with GPs and one with pairs.

SECONDARY OUTCOMES:
Acceptability 1 | 3 months after last inclusion
  Number of clusters included / Number of clusters planned measured by logbooks
Acceptability 2 | within 6 months after refusal
  Reason for pharmacists and general practitioners' refusal assesed by individual interviews
Acceptability 3 | 3 months after last inclusion
  Number of patients included / Number of patients eligible measured by logbooks
Cost-Utility analysis assessed following the Haute Autorité de Santé 2020 recommendations | 12 months after the last inclusion
  A Cost-Utility Analysis (CUA) expressed as a cost per Quality Adjusted Life Year (QALY) will be performed from a collective perspective and with a time horizon of 12 months
Fidelity 1 | 12 months after the last inclusion
  Proportion of pairs completing the study measured through a logbook
Fidelity 2 | 12 months after the last inclusion
  Proportion of patients who actually made appointments with the pharmacist measured through a logbook.
Fidelity 3 | 6 months after the last inclusion
  Number of motivational interviews measured through a logbook.
Fidelity 4 | 6 months after the last inclusion
  Number of reporting made by the pharmacist to the GP will be measured through a logbook.
BZDR consumption | 10 to 12 months after enrollment in the study
  Cessation or reduction of BZDR use at 12 months from inclusion measured using the National Health Data System.
  Proportion of patients no longer being dispensed BZDR at 10 months after enrollment, with the last two months (10 to 12 months)
Anxiety | 6 and 12 months after enrollment
  Anxiety measured by General Anxiety Disorder (GAD-7)
Insomnia | 6 and 12 months after enrollment
  Quality of sleep measured by Insomnia Severity Index (ISI)
Attachment to BZDR | 6 and 12 months after enrollment
  Attachment to BZDR measured by Benzodiazepine Cognitive Attachment Scale (ECAB) scale at 6 and 12 months.
  Score ranges from 0 to 10. A score ≥ 6 allows
Reported Quality of life of patients | 6 and 12 months after enrollment
  Quality of life measured by EQ-5D-5L questionnaire at 6 and 12 months. A total of 3125 possible health states is defined. Each state is referred to by a 5-digit code.
Autonomy | 6 and 12 months after enrollment
  Autonomy measured by Instrumental Activities of Daily Living (IADL) at 6 and 12 months.
  The scale ranges from 0 to 8, with 0 indicating complete dysautonomia and 8 indicating complete autonomy.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-François HUON, Pharm.D PhD, Principal Investigator — Nantes University Hospital

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Huon JF, Nizet P, Caillet P, Lecompte H, Victorri-Vigneau C, Fournier JP; BESTOPH-MG consortium. Evaluation of the effectiveness of a joint general practitioner-pharmacist intervention on the implementation of benzodiazepine deprescribing in older adults (BESTOPH-MG trial): protocol for a cluster-randomized controlled trial. Front Med (Lausanne). 2023 Aug 25;10:1228883. doi: 10.3389/fmed.2023.1228883. eCollection 2023. PMID 37711743